CLINICAL TRIAL: NCT00134966
Title: A 39 Week Randomized, Double-Blind, Parallel Group, Multicenter Study to Evaluate the Effect of Fixed Dose Carbidopa/Levodopa/Entacapone 100 mg t.i.d. vs. Immediate Release Carbidopa/Levodopa 25/100 mg (t.i.d.) in Parkinson's Disease Patients Requiring Levodopa
Brief Title: A Study to Evaluate Fixed Dose Carbidopa/Levodopa/Entacapone Versus Immediate Release Carbidopa/Levodopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CELC200A2305
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease, levodopa, dyskinesia
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Levodopa; entacapone; Stalevo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: capsules containing: carbidopa (25 mg), levodopa (100 mg), entacapone (200 mg)
- 2 (Active Comparator)
  Interventions: Drug: capsules containing: carbidopa (25 mg), levodopa (100 mg), entacapone (200 mg)

INTERVENTIONS:
Drug: capsules containing: carbidopa (25 mg), levodopa (100 mg), entacapone (200 mg)
  Other Names: Stalevo; CELC200

SUMMARY:
The purpose of this study is to achieve approval for the use of carbidopa/levodopa/entacapone in early Parkinson's disease (PD) by demonstrating that when used as initial levodopa therapy in early PD, carbidopa/levodopa/entacapone provides significantly greater symptomatic benefit than immediate release carbidopa/levodopa administered at the same levodopa dosage level of 100 mg three times a day (t.i.d.).

DETAILED DESCRIPTION:
The purpose of this study is to achieve approval for the use of carbidopa/levodopa/entacapone in early Parkinson's disease (PD) by demonstrating that when used as initial levodopa therapy in early PD, carbidopa/levodopa/entacapone provides significantly greater symptomatic benefit than immediate release carbidopa/levodopa administered at the same levodopa dosage level 100 mg t.i.d.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 to 80 years, inclusive, at time of Parkinson's disease diagnosis
* Idiopathic Parkinson's disease with at least 2 cardinal signs of disease: resting tremor, bradykinesia or rigidity
* Parkinson's disease impairment warranting treatment with a levodopa formulation according to the investigator's assessment

Exclusion Criteria:

* History, signs or symptoms suggesting the diagnosis of atypical or secondary Parkinsonism due to drugs, metabolic disorders, encephalitis or other neurodegenerative diseases
* History of stereotaxic brain surgery for PD (e.g., pallidotomy, deep brain stimulation, tissue transplant)
* Diagnosis of Parkinson's disease for more than 5 years prior to Screening
* Previous use of levodopa in any formulation, entacapone or tolcapone for more than 30 days or anytime within 4 weeks (28 days) prior to baseline
* Use of a dopamine agonist within 4 weeks (28 days) prior to baseline

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2005-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Symptom control change from baseline to week 39

SECONDARY OUTCOMES:
Change from baseline to week 39 in activities of daily living
Change from baseline to week 39 in motor function
Change from baseline to week 39 in mental acuity
Change from baseline to week 39 in incidence of dyskinesia and wearing off

CONTACTS AND LOCATIONS:
Locations (60):
- United States (17):
  - Barrow Neurology Clinics at St. Joseph's Hosptial & Medical Center, Phoenix, Arizona
  - Coastal Neurological Medical Group, Inc, La Jolla, California
  - Neurosearch, Inc., Reseda, California
  - University of Florida Health Science Center, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - USF Medical Clinic, Tampa, Florida
  - Springfield Neurology Associates, LLC, Springfield, Massachusetts
  - Clinical Neuroscience Center, Southfield, Michigan
  - Melbourne Internal Medicine Associates, Westlake, Ohio
  - Westmoreland Neurology Associates, Inc., Greensburg, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - NeuroHealth, Warwick, Rhode Island
  - Coastal Neurology, PA, Beaufort, South Carolina
  - Senior Adults Specialty Research, Austin, Texas
  - Baylor College of Medicine, Parkinson's Disease Center, Houston, Texas
  - Neurology Associates, San Marcos, Texas
  - Blue Ridge Research Center at Roanoke Neurological Center, Roanoke, Virginia
- Canada (18):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - Moncton, New Brunswick
  - Eastern Health Care - Health Sciences Centre, Neurology Department, HSC Room 5317, 300 Prince Philip Drive, Saint John's, Newfoundland and Labrador
  - Neurology Division, Health Science Center, Halifax, Nova Scotia
  - Cape Breton Regional Hospital, Neurology Department, Sydney, Nova Scotia
  - Grand River Hospital, Kitchener, Ontario
  - London Health Sciences Center, University Hospital, Rm. A10-026, London, Ontario
  - Centre for Movement Disorders, Markham, Ontario
  - Parkinson's & Neurodegenerative Disorders Clinic, Ottawa, Ontario
  - Ottawa Hospital, Civic Campus, Ottawa, Ontario
  - Hiren Desai Medicine Professional Corporation, Windsor, Ontario
  - Neuro Rive Sud, Greenfield Park, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Unite des Troubles du Mouvement Andre-Barbeau, CHUM-Hotel-Dieu, Montreal, Quebec
  - Centre de Recjerche Clinique du CHUS, Sherbrooke, Quebec
  - Dr. Felix Veloso Research, Regina, Saskatchewan
  - Quebec Memory and Motor Skills Disorders Clinic, Québec
  - University of Saskatchewan, Royal University Hospital, Saskatoon
- Czechia (4):
  - Neurologická klinika, Univerzita Palackého, I.P.Pavlova 6, Olomouc
  - FN-neurologická klinika, Alej Svobody 80, Plzeň
  - Neurologicka klinika, Katerinska 12, Praha 2
  - FN-Nemocnice Pardubice, Kyjevska 44, Pardubice
- Israel (4):
  - Rambam Medical Center, Haliya Hashniya 8, Haifa District
  - Dep. Of Neurology (Bitan 38, EEG institute), Dep. of Neurology, Zerifin
  - Belinson Campus, Jabotinsky st. Movement Disorder Unit, Petah Tikva
  - Sourasky Medical Center, Weitzman Saint Movement Disorder Clinic, Tel Aviv
- Italy (8):
  - Clinica Neurologica I - Azienda Ospedaliera-Universitaria Policlinico - Università di Catania, Via Santa Sofia 78, Catania
  - "Dipartimento di Neuroscienze Oftalmologia e Genetica (DINOG), Università Degli Studi Di Genova, Via de Toni 5, Genova
  - Unità Operativa Complessa Neurologia - Policlinico Universitario "G. Martino", Via Consolare Valeria, Messina
  - Istituto Nazionale Neurologico "Carlo Besta", Via Celoria 11, Milano
  - Dipartimento di Neuroscienze-Sezione Neurologia Università degli Studi di Pisa- AO S. Chiara, Via Roma, 67, Pisa
  - Dipartimento di Scienze Neurologiche Università degli Studi di Roma "La Sapienza" Roma I, Viale dell'Università 30, Roma
  - Dipartimento di Neuroscienze-Università degli Studi di Torino, Via Cherasco 15, Torino
  - A.O. Istituti Clinici di Perfezionamento-Unita'Operativa Centro Parkinson, Via Bignami 1, Milan
- Poland (3):
  - Samodzielny Publiczny Szpital Kliniczny Oddzial Kliniczny Neurologii i Epiletologii, Ul. Czerniakowska 231, Warszawa
  - Centrum Neurologii Klinicznej, Ul. Dwernickiego 8, Krakow
  - Klinika Neruologii Wieku Podeszlego, ul.Medykow 14, Katowice
- Portugal (3):
  - Hospitais da Universidade de Coimbra (Serv. Neurologia), Avenida Bissaya Barreto, Coimbra
  - Hospital de Santa Maria (Serv. Neurologia), Avenida Professor Egas Moniz, Lisbon
  - Hospital de Santo António (Serv. Neurologia), Largo Professor Abel Salazar, Porto
- Turkey (Türkiye) (3):
  - Istanbul CAPA Medical School, Istanbul University CAPA Medical School, Dept. of Neurology, Istanbul
  - Hacettepe Medical School, Department of Neurology, Hacettepe Universitesi Hastaneleri Norooji AD Sihhiye, Ankara
  - Dokuz Eylul Medical School, Department of Neurology, Noroloji Anabilim Dali Inciralti Izmir, Izmir

REFERENCES:
- [Derived] Hauser RA, Panisset M, Abbruzzese G, Mancione L, Dronamraju N, Kakarieka A; FIRST-STEP Study Group. Double-blind trial of levodopa/carbidopa/entacapone versus levodopa/carbidopa in early Parkinson's disease. Mov Disord. 2009 Mar 15;24(4):541-50. doi: 10.1002/mds.22343. PMID 19058133